CLINICAL TRIAL: NCT04675710
Title: Pembrolizumab in Combination With Dabrafenib and Trametinib as a Neoadjuvant Strategy Prior to Surgery in BRAF-Mutated Anaplastic Thyroid Cancer
Brief Title: Pembrolizumab, Dabrafenib, and Trametinib Before Surgery for the Treatment of BRAF-Mutated Anaplastic Thyroid Cancer
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2020-0641; NCI-2020-09803 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2020-0641 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2020-12-05; First posted 2020-12-19 (Actual); Last update posted 2025-10-14 (Actual); Status verified 2025-08

CONDITIONS: Thyroid Gland Anaplastic Carcinoma; Thyroid Gland Squamous Cell Carcinoma
MeSH Terms: conditions — Thyroid Carcinoma, Anaplastic | interventions — dabrafenib; Radiotherapy, Intensity-Modulated; pembrolizumab; trametinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (dabrafenib, trametinib, pembrolizumab) (Experimental): Patients receive 21-day cycles of dabrafenib 150 mg orally (PO) twice daily from Days 1-21, trametinib 2mg PO once daily from Days 1-21, and pembrolizumab 200mg intravenously (IV) on Day 1 of each cycle.
  Interventions: Procedure: Conventional Surgery; Drug: Dabrafenib; Radiation: Intensity-Modulated Radiation Therapy; Biological: Pembrolizumab; Other: Quality-of-Life Assessment; Drug: Trametinib

INTERVENTIONS:
Procedure: Conventional Surgery — Undergo surgery
Drug: Dabrafenib — Given PO
  Other Names: BRAF Inhibitor GSK2118436; GSK-2118436; GSK-2118436A; GSK2118436
Radiation: Intensity-Modulated Radiation Therapy — Undergo IMRT
  Other Names: IMRT; Intensity Modulated RT; Intensity-Modulated Radiotherapy; Radiation, Intensity-Modulated Radiotherapy
Biological: Pembrolizumab — Given IV
  Other Names: Keytruda; Lambrolizumab; MK-3475; SCH 900475
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Drug: Trametinib — Given PO
  Other Names: GSK1120212; JTP-74057; MEK Inhibitor GSK1120212; Mekinist

SUMMARY:
This phase II trial studies the effect of pembrolizumab, dabrafenib, and trametinib before surgery in treating patients with BRAF V600E-mutated anaplastic thyroid cancer. BRAF V600E is a specific mutation (change) in the BRAF gene, which makes a protein that is involved in sending signals in cells and in cell growth. It may increase the growth and spread of tumor cells. Dabrafenib and trametinib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Immunotherapy with monoclonal antibodies, such as pembrolizumab, may help the body's immune system attack the cancer, and may interfere with the ability of tumor cells to grow and spread. Pembrolizumab, dabrafenib, and trametinib may help to control BRAF V600E-mutated anaplastic thyroid cancer when given before surgery.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Demonstrate the efficacy of upfront treatment with neoadjuvant pembrolizumab in combination dabrafenib and trametinib by comparing the complete gross surgical resection rate (R0 or R1 surgical resection) to historical control of 5%.

II. Demonstrate the efficacy of pembrolizumab in combination with dabrafenib and trametinib by comparing the overall survival (OS) to historical OS rate of 9.6 months.

SECONDARY OBJECTIVES:

I. Assess the efficacy (Response Evaluation Criteria in Solid Tumors [RECIST]) of neoadjuvant dabrafenib, trametinib, and pembrolizumab combination (Part 1) and progression-free survival (PFS) for all patients throughout their treatment course.

II. Demonstrate the extent to which neoadjuvant dabrafenib, trametinib, and pembrolizumab changes surgical morbidity/complexity.

III. Establish surgical safety for neoadjuvant pembrolizumab in combination with BRAF & MEK inhibitors, dabrafenib and trametinib; as well as safety for concurrent administration of postoperative adjuvant pembrolizumab with intensity modulated radiation therapy (IMRT).

VI. Evaluate changes in patient reported outcomes: quality of life assessed by validated questionnaires at initial diagnosis, through the course of therapy, and during the adjuvant targeted therapy phase.

VII. Determine whether features of the tumor genomic landscape and tumor immune microenvironment are associated with response to dabrafenib/trametinib/pembrolizumab (DTP).

EXPLORATORY OBJECTIVES:

I. Determine if changes of cell free deoxyribonucleic acid (DNA) correlate with response to treatment on DTP and overall survival.

II. Evaluate the safety of dabrafenib/trametinib/pembrolizumab plus IMRT in a subset of 15 patients.

OUTLINE:

PART 1 (NEOADJUVANT PHASE): Patients receive dabrafenib orally (PO) twice daily (BID) and trametinib PO once daily (QD) on days 1-21. Starting in week 4, patients also receive pembrolizumab intravenously (IV) over 30 minutes on day 1. Treatment repeats every 21 days for 3 cycles in the absence of disease progression or unacceptable toxicity. Patients may receive 2 additional cycles of DTP at the discretion of the treating physicians. Patients whose disease is deemed resectable undergo surgery. Patients who are not surgically resectable after 5 cycles of DTP move to Part 3.

PART 2 (ADJUVANT PHASE): 2-4 weeks after surgery and at the discretion of the treating physicians, patients may continue to receive pembrolizumab IV over 30 minutes every 3 weeks and concurrently undergo IMRT with or without cisplatin or carboplatin for 6 weeks. Up to 15 patients also receive dabrafenib PO BID and trametinib PO QD concurrently for 6 weeks.

PART 3: Patients receive dabrafenib PO BID, trametinib PO QD on days 1-21, and pembrolizumab IV over 30 minutes on day 1. Treatment repeats every 21 days for 17 cycles in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 3 months during years 1-2, every 6 months during years 3-4, and then annually thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Pathologic findings supporting the clinical impression of anaplastic thyroid carcinoma. Diagnosis may include consistent with or suggestive of terminology associated with: anaplastic thyroid carcinoma, undifferentiated carcinoma, squamous carcinoma; carcinoma with spindled, giant cell, or epithelial features; poorly differentiated carcinoma with pleomorphism, extensive necrosis with tumor cells present
* Must have a BRAFV600E mutation-positive tumor, as determined by BRAF V600E immunohistochemistry on tumor tissue, genetic/molecular testing of tumor, or cell free (cf)NDA liquid biopsy
* Have measurable disease based on RECIST 1.1
* Total bilirubin =< 1.5 x upper limit of normal (ULN). Total bilirubin =< 3 x ULN for patients with Gilbert's syndrome
* Aspartate aminotransferase (AST) (serum glutamic-oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 2.5 x ULN, (5 x ULN for patients with concurrent liver metastases)
* Serum creatinine =< within 1.5 x ULN
* Absolute neutrophil count (ANC) >= 1.0 x 10^9/L
* Platelets >= 100 x 10^9/L
* Hemoglobin >= 9.0 g/dL or 5.6 mmol/L
* International normalized ratio (INR) or prothrombin time (PT) =< 1.5 x ULN unless participant is receiving anticoagulant therapy as long as PT or activated partial thromboplastin time (aPTT) is within therapeutic range of intended use of anticoagulant
* Subjects must be willing to ultimately undergo surgery if their tumor becomes surgically resectable. For MD Anderson site only, subjects must be willing to undergo tumor biopsy after the run-in with DT, unless in the opinion of the treating physician, a biopsy is not feasible or safe. Research subjects retain the right to refuse any research interventions.
* Have an Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1. Evaluation of ECOG is to be performed within 7 days prior to the date of allocation/randomization
* The participant (or legally acceptable representative if applicable) provides written informed consent for the trial
* A male participant must agree to use a contraception of this protocol during the treatment period and for at least 8 months after the last dose of study treatment and refrain from donating sperm during this period
* A female participant is eligible to participate if she is not pregnant, not breastfeeding, and at least one of the following conditions applies:

  * Not a woman of childbearing potential (WOCBP) OR
  * A WOCBP who agrees to follow the contraceptive guidance during the treatment period and for at least 6 months after the last dose of study treatment

Exclusion Criteria:

* Significant cardiovascular impairment: history of congestive heart failure greater than New York Heart Association (NYHA) class II
* Untreated brain metastases
* Prior chemotherapy within < 1 week prior to study day 1 or patients who have not recovered (i.e., =< grade 2) from adverse events due to a previously administered agent, except for patients who have been on dabrafenib/trametinib (DT) according to the standard run-in outlined in the trial schema
* Has active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment
* History of human immunodeficiency virus (HIV) or active hepatitis B (chronic or acute) or hepatitis C infection. Patients with past or resolved hepatitis B infection (defined as having a negative hepatitis B surface antigen [HBsAg] test and a positive anti-HBc [antibody to hepatitis B core antigen] antibody test) are eligible. However, patients with past or resolved hepatitis B virus (HBV) should be monitored for reactivation by a specialist. Patients positive for hepatitis C virus (HCV) antibody are eligible only if polymerase chain reaction (PCR) is negative for HCV ribonucleic acid (RNA). Note: no testing for HIV, hepatitis B and hepatitis C is required unless mandated by local heath authority
* Has a diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy (in dosing exceeding 10 mg daily of prednisone equivalent) or any other form of immunosuppressive therapy within 7 days prior to the first dose of study drug
* Has received a live or live-attenuated vaccine within 30 days prior to the first dose of study drug. Administration of killed vaccines is allowed
* Has severe hypersensitivity (>= grade 3) to pembrolizumab and/or any of its excipients
* Has a history of (non-infectious) pneumonitis/interstitial lung disease that required steroids or has current pneumonitis/interstitial lung disease
* Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial
* Females who are breastfeeding or pregnant at screening or baseline (as documented by a positive beta-human chorionic gonadotropin [beta-hCG] (or human chorionic gonadotropin [hCG]) test with a minimum sensitivity of 25 IU/L or equivalent units of beta-hCG [or hCG]). A women of childbirth potential (WOCBP) who has a positive urine pregnancy test within 72 hours prior to the first infusion will be excluded. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required
* More than 42 days of DT therapy prior to enrollment
* A known history of retinal vein occlusion (RVO), central serous retinopathy (CSR), uncontrolled glaucoma or ocular hypertension

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-06-24 (Actual); Primary Completion 2026-10-30 (Estimated); Study Completion 2026-10-30 (Estimated)

PRIMARY OUTCOMES:
Complete gross surgical resection (R0 or R1 resection) | Up to 5 cycles (1 cycle = 21 days) Up to 7 cycles
  Overall R0/R1 resection rate will be defined by proportion of patients who undergo successful thyroidectomy with clear (R0) or microscopically positive (R1) surgical margins. We will test the hypothesis that the R0/R1 resection rate is greater than historical rate of 5%.
Overall survival (OS) | Up to 72 months
  OS will be measured as the time from the start of any trial treatment to death from any causes. Kaplan-Meier method will be used to estimate the median survival time across all patients and its 95% confidence intervals (CI).

SECONDARY OUTCOMES:
Tumor response | Up to 42 months
  Objective tumor response will be assessed by Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1.
Progression free survival (PFS) | Up to 42 months
  PFS will be measured as the time from the start of the treatment to the first occurrence of disease progression or death from any cause, whichever occurs first, as determined by RECIST version 1.1.
Surgical morbidity/complexity | Up to 5 cycles (1 cycle = 21 days) Up to 7 cycles
  Surgical morbidity/complexity will be measured at enrollment, prior to surgery and at surgery. The Thyroid Neck Group Morbidity Complexity Scoring and MGH/MEE-MSK-MD Anderson (MMM) Surgical Morbidity Complexity Score are incorporated, specifying on a scale with 5 levels of complexity and morbidity of the surgery [mild (level 0), moderate (level 1), severe (level 2), very severe (level 3), and unresectable (level 4)].
Number of patients with adverse events as a measure of safety of neoadjuvant dabrafenib, trametinib, and pembrolizumab | Up to 5 cycles (1 cycle = 21 days)
  Frequency and severity of adverse events as a measure of safety profile for neoadjuvant concurrent administration of dabrafenib, trametinib, and pembrolizumab (DTP) will be assessed using Common Terminology Criteria for Adverse Events version 5.0.
Number of patients with adverse events as a measure of safety of postoperative pembrolizumab plus IMRT | Over the course of adjuvant IMRT plus 2 weeks of safety follow-up, assessed up to 2 months
  Frequency and severity of adverse events as a measure of safety profile for concurrent administration of postoperative pembrolizumab with IMRT will be assessed using Common Terminology Criteria for Adverse Events version 5.0.
Locoregional control | Up to 42 months
  Locoregional control will be measured as the time from the start of any trial treatment to the first locoregional recurrence/progression event.
Health related quality of life | Up to 42 months
  Changes of health-related quality of life will be measured by the European Quality of Life 5 Dimension Questionnaire (EQ-5D). The EQ-5D consists of health state description and evaluation. The health state description consists of five dimensions (mobility, self-care, usual activities, pain/discomfort, and anxiety/depression), with each dimension specifying five levels of severity [best (1)-worst (5)]. The health state evaluation is assessed using the visual analogue scale ([worse (0)-best (100)].
Patient-reported symptoms | Up to 42 months
  Symptom burden experienced by patients will be measured by the M.D. Anderson Symptom Inventory for Head and Neck Cancer (MDASI-HN) instrument.

CONTACTS AND LOCATIONS:
Overall Officials: Mark Zafereo, Principal Investigator — M.D. Anderson Cancer Center
Locations (6):
- United States (6):
  - Stanford School of Medicine, Stanford, California
  - University of Michigan Rogel Cancer Center, Ann Arbor, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - Cleveland Clinic Taussig Cancer Institute, Cleveland, Ohio
  - M D Anderson Cancer Center, Houston, Texas
  - Huntsman Cancer Institute at the University of Utah, Salt Lake City, Utah

REFERENCES:
- See also: MD Anderson Cancer Center — http://www.mdanderson.org